CLINICAL TRIAL: NCT01746901
Title: A Randomized, Double-blind, Double-dummy, Placebo Controlled, Single-dose, 6-way Crossover Study To Determine The Relative Abuse Potential Of Alo-02 (Oxycodone Hydrochloride And Naltrexone Hydrochloride Extended-release Capsules) Compared To Oxycodone Immediate Release And Placebo When Administered Orally To Nondependent,Recreational Opioid Users.
Brief Title: A Study to Characterize the Abuse Liability of ALO-02 in Healthy, Non-Dependent, Recreational Opioid Abusers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: B4531008
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Relative abuse potential study; oxycodone; nalteone; Opioid-related disorders; drug abusers; Chronic pain
MeSH Terms: conditions — Opioid-Related Disorders; Drug Misuse; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment B (Experimental)
  Interventions: Drug: intact ALO-02 60 mg/7.2 mg
- Treatment C (Experimental)
  Interventions: Drug: crushed ALO-02 60 mg/7.2 mg
- Treatment D (Active Comparator)
  Interventions: Drug: crushed oxycodone IR 60 mg
- Treatment E (Experimental)
  Interventions: Drug: crushed ALO-02 40 mg/4.8 mg
- Treatment F (Active Comparator)
  Interventions: Drug: crushed oxycodone IR 40 mg

INTERVENTIONS:
Drug: Placebo — Placebo solution + Placebo ALO-02 (intact)
  Arms: Treatment A
Drug: intact ALO-02 60 mg/7.2 mg — Placebo solution + ALO-02 60 mg/7.2 mg (intact)
  Arms: Treatment B
Drug: crushed ALO-02 60 mg/7.2 mg — crushed ALO-02 60 mg/7.2 mg in solution + placebo ALO-02 (intact)
  Arms: Treatment C
Drug: crushed oxycodone IR 60 mg — crushed oxycodone immediate-release (IR) 60 mg in solution + placebo ALO-02 (intact)
  Arms: Treatment D
Drug: crushed ALO-02 40 mg/4.8 mg — crushed ALO-02 40 mg/4.8 mg in solution + placebo ALO-02 (intact)
  Arms: Treatment E
Drug: crushed oxycodone IR 40 mg — crushed oxycodone immediate-release (IR) 40 mg in solution + placebo ALO-02 (intact)
  Arms: Treatment F

SUMMARY:
The main purpose of this study is to determine if oxycodone and naltrexone combination capsules (ALO-02) have the potential to be abused.

DETAILED DESCRIPTION:
Abuse Liability Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects.
* Non-dependent, recreational opioid users. (Must use opioid for non-therapeutic purposes on at least 10 occassions within the last year before Screening Visit, and at least once in 8 weeks before the Screening Visit.

Exclusion Criteria:

* Diagnosis of substance and/or alcohol dependence.
* Subject has participated in, is currently participating in, or is seeking treatment for substance and/or alcohol related disorder.
* History of sleep apnea.
* Positive urine drug screen (UDS) for other that marijuana.
* Positive for Hepatitis B or C and HIV on Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- INC Research Toronto, Inc., Toronto, Ontario, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531008&StudyName=A%20Study%20to%20Characterize%20the%20Abuse%20Liability%20of%20ALO-02%20in%20Healthy%2C%20Non-Dependent%2C%20Recreational%20Opioid%20Abusers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recreational opioid users who were not dependent on opioids based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR) criteria, were recruited in this study.
Pre-assignment Details: After successful naloxone challenge test, all participants underwent training sessions involving complete pharmacodynamics test battery before the drug discrimination phase, to ensure that participants fully understood how to perform the tests, were comfortable, and attained a stable level of performance on the various performance-based measures.
Groups:
- Naloxone: Naloxone hydrochloride (HCl) 0.2 milligram (mg) intravenously followed by additional 0.6 mg naloxone hydrochloride intravenously on Day 0, each dose followed by an assessment for signs and symptoms of opioid withdrawal. Participants who did not display signs and symptoms of opioid withdrawal, were assigned to either oxycodone HCl 40 mg then placebo or placebo then oxycodone HCl 40 mg group in the drug discrimination phase of the study.
- Oxycodone HCl 40 mg Then PBO: Single dose of oxycodone HCl 40 mg crushed tablet in solution, orally on Day 1 followed by single dose of placebo matched to oxycodone HCl crushed tablet orally on Day 2. Participants were assigned to receive oxycodone HCl 60 mg and naltrexone HCl 7.2 mg extended-release (ALO-02) 60 mg/7.2 mg intact capsule, ALO-02 60 mg/7.2 mg and ALO-02 40 mg/4.8 mg crushed capsule in solution, oxycodone HCl 40 mg (OXY 40 mg) and 60 mg crushed tablet (OXY 60 mg) in solution, placebo matched to either ALO-02 intact (PBO) and crushed capsule or oxycodone crushed tablet (PBO), orally, in either of the 6 sequences in the treatment phase of the study.
- PBO Then Oxycodone HCl 40 mg: Single dose of placebo matched to oxycodone HCl crushed tablet orally on Day 1 followed by single dose of oxycodone HCl 40 mg crushed tablet in solution, orally on Day 2. Participants were assigned to receive oxycodone HCl 60 mg and naltrexone HCl 7.2 mg extended-release (ALO-02) 60 mg/7.2 mg intact capsule, ALO-02 60 mg/7.2 mg and ALO-02 40 mg/4.8 mg crushed capsule in solution, oxycodone HCl 40 mg (OXY 40 mg) and 60 mg crushed tablet (OXY 60 mg) in solution, placebo matched to either ALO-02 intact (PBO) and crushed capsule or oxycodone crushed tablet (PBO), orally, in either of the 6 sequences in the treatment phase of the study.
- ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C: Single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in first intervention period; followed by single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in second intervention period; then single dose of matching placebo (PBO) orally on Day 1 in third intervention period; then single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in fourth intervention period; then single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on Day 1 in fifth intervention period; then single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I: Single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally on Day 1 in first intervention period; followed by single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on orally on Day 1 in second intervention period; then single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in third intervention period; then single dose of matching placebo (PBO) orally on Day 1 in fourth intervention period; then single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in fifth intervention period; then single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg: Single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in first intervention period; followed by single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in second intervention period; then single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in third intervention period; then single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally on Day 1 in fourth intervention period; then single dose of matching placebo (PBO) orally on Day 1 in fifth intervention period; then single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C: Single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on Day 1 in first intervention period; followed by single dose of matching placebo (PBO) orally on Day 1 in second intervention period; then single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally on Day 1 in third intervention period; then single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in fourth intervention period; then single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in fifth intervention period; then single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO: Single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in first intervention period; followed by single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally on Day 1 in second intervention period; then single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in third intervention period; then single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on Day 1 in fourth intervention period; then single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in fifth intervention period; then by single dose of matching placebo (PBO) orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg: Single dose of matching placebo (PBO) orally on Day 1 in first intervention period; followed by single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally on Day 1 in second intervention period; then single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally on Day 1 in third intervention period; then single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally on Day 1 in fourth intervention period; then single dose of ALO-02 40 mg/4.8 mg crushed capsule (ALO-02 40 mg-I) solution orally on Day 1 in fifth intervention period; then single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally on Day 1 in sixth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
Period: Naloxone Challenge Phase
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 75 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 72 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet entrance criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 1
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 33 | 36 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 2
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 33 | 36 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 19 | 22 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 14 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not met entrance criteria | 0 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: First Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 7 | 8 | 7 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Phase: Washout Period 1
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 7 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Second Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 7 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Phase: Washout Period 2
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 6 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Third Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 7 | 7 | 6 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Period: Treatment Phase: Washout Period 3
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 7
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Fourth Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 7
Completed | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Period: Treatment Phase: Washout Period 4
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Completed | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Fifth Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Completed | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period 5
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Completed | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Sixth Intervention
Arm/Group | Naloxone | Oxycodone HCl 40 mg Then PBO | PBO Then Oxycodone HCl 40 mg | ALO-02 60 Mg-I,ALO-02 60 Mg-C,PBO,OXY 60,40 mg,ALO-02 40 Mg-C | ALO-02 40 Mg-C,OXY 40,60 mg,PBO,ALO-02 60 Mg-C,ALO-02 60 Mg-I | ALO-02 60 Mg-C,OXY 60 mg,ALO-02 60 Mg-I,40 Mg-C,PBO,OXY40 mg | OXY 40 mg,PBO,ALO-02 40 Mg-C,60 Mg-I,OXY 60 mg,ALO-02 60 Mg-C | OXY 60 mg,ALO-02 40, 60 Mg-C,OXY 40 mg,ALO-02 60 Mg-I,PBO | PBO,ALO-02 60 Mg-I,OXY 40 mg, ALO-02 60, 40 Mg-C,OXY 60 mg
Started | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Completed | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Entire Study Population: Included all participants enrolled in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking: Peak Effect (Emax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the extreme left with "strong disliking" (score of 0 mm) and on the extreme right with "strong liking" (score of 100 mm). Peak Effect (Emax) = Maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose in treatment phase
Population: Completer analysis set included all randomized participants who completed all 6 periods of treatment phase and who contributed to post-dose Pharmacodynamic (PD) data from each period.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo: Single dose of matching placebo solution orally in either of the first to sixth intervention periods.
- ALO-02 40 Mg-C: Single dose of ALO-02 40 mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally in either of the first to sixth intervention periods.
- OXY 40 mg: Single dose of oxycodone HCl 40 mg (OXY 40 mg) crushed tablet solution orally in either of the first to sixth intervention periods.
- ALO-02 60 Mg-I: Single dose of ALO-02 60 mg/7.2 mg intact capsule (ALO-02 60 mg-I) solution orally in either of the first to sixth intervention periods.
- ALO-02 60 mg- C: Single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally in either of the first to sixth intervention periods.
- OXY 60 mg: Single dose of oxycodone HCl 60 mg (OXY 60 mg) crushed tablet solution orally in either of the first to sixth intervention periods.
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 51.6 (3.74) | 70.1 (19.23) | 85.5 (16.11) | 59.3 (15.09) | 74.4 (18.10) | 89.7 (13.59)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least Squares (LS) Mean Difference = 30.5, 95% CI 2-sided [24.4 to 36.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0132, Mixed Models Analysis; LS Mean Difference = 7.7, 95% CI 2-sided [1.6 to 13.7]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 15.3, 95% CI 2-sided [9.3 to 21.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 22.9, 95% CI 2-sided [16.8 to 28.9]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 15.3, 95% CI 2-sided [9.3 to 21.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 18.5, Mixed Models Analysis; LS Mean Difference = 18.5, 95% CI 2-sided [12.5 to 24.6]

2. Primary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-2 Hour
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the extreme left with "strong disliking" (score of 0 mm) and on the extreme right with "strong liking" (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hours.
Time Frame: 0.25, 0.5, 1, 1.5, 2 hours post-dose
Population: Completer analysis set included all randomized participants who completed all 6 periods of treatment phase and who contributed to post-dose PD data from each period.
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm | 100.004 (5.1468) | 118.480 (28.7707) | 141.305 (32.9203) | 100.188 (10.6437) | 127.320 (31.2906) | 149.484 (24.1907)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 49.3, 95% CI 2-sided [39.2 to 59.5]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9994, Mixed Models Analysis; LS Mean Difference = 0.0, 95% CI 2-sided [-10.1 to 10.1]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 22.2, 95% CI 2-sided [12.1 to 32.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 27.1, 95% CI 2-sided [17.0 to 37.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 23.0, 95% CI 2-sided [12.8 to 33.1]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; LS Mean Difference = 18.2, 95% CI 2-sided [8.1 to 28.4]

3. Primary Outcome: High: Peak Effect (Emax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose in treatment phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 10.9 (20.60) | 47.3 (36.88) | 77.9 (25.46) | 21.7 (35.36) | 53.4 (34.68) | 84.7 (23.67)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 63.2, 95% CI 2-sided [51.5 to 74.9]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0402, Mixed Models Analysis; LS Mean Difference = 12.3, 95% CI 2-sided [0.6 to 24.1]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 32.9, 95% CI 2-sided [21.1 to 44.7]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 42.6, 95% CI 2-sided [30.9 to 54.4]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 32.1, 95% CI 2-sided [20.3 to 43.9]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 36.3, 95% CI 2-sided [24.6 to 48.1]

4. Primary Outcome: High: Area Under Effect Curve (AUE) From 0-2 Hour
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hours.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm | 2.496 (8.3003) | 55.250 (54.1280) | 112.082 (43.7000) | 9.902 (21.1911) | 71.254 (55.9812) | 117.578 (42.2152)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 108.0, 95% CI 2-sided [91.6 to 124.5]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4125, Mixed Models Analysis; LS Mean Difference = 6.8, 95% CI 2-sided [-9.6 to 23.3]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 46.1, 95% CI 2-sided [29.6 to 62.5]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 68.8, 95% CI 2-sided [52.4 to 85.2]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 56.7, 95% CI 2-sided [40.3 to 73.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 52.6, 95% CI 2-sided [36.2 to 69.0]

5. Secondary Outcome: Take Drug Again: Peak Effect (Emax)
Description: Take drug again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely would not", 50 mm = "do not care", and 100 mm = "definitely would"). Emax = Maximum observed score.
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 45.7 (19.05) | 57.9 (33.58) | 83.4 (20.26) | 48.1 (28.14) | 72.0 (28.31) | 81.3 (25.23)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 32.8, 95% CI 2-sided [21.8 to 43.7]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6434, Mixed Models Analysis; LS Mean Difference = 2.6, 95% CI 2-sided [-8.4 to 13.5]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1072, Mixed Models Analysis; LS Mean Difference = 9.0, 95% CI 2-sided [-2.0 to 20.0]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.3, 95% CI 2-sided [15.4 to 37.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.7, 95% CI 2-sided [14.7 to 36.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0335, Mixed Models Analysis; LS Mean Difference = 11.9, 95% CI 2-sided [0.9 to 22.9]

6. Secondary Outcome: Take Drug Again: Mean Effect (Emean)
Description: as for outcome 5
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 42.90 (20.002) | 54.71 (32.635) | 77.80 (22.880) | 42.63 (26.293) | 68.78 (29.883) | 78.02 (24.868)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 35.0, 95% CI 2-sided [24.0 to 46.0]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9811, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-11.1 to 10.8]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1083, Mixed Models Analysis; LS Mean Difference = 9.0, 95% CI 2-sided [-2.0 to 19.9]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.9, 95% CI 2-sided [14.9 to 36.9]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 23.2, 95% CI 2-sided [12.3 to 34.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0408, Mixed Models Analysis; LS Mean Difference = 11.5, 95% CI 2-sided [0.5 to 22.4]

7. Secondary Outcome: Take Drug Again: Minimum Effect (Emin)
Description: as for outcome 5
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 41.1 (21.60) | 50.9 (32.46) | 73.2 (26.92) | 37.8 (28.72) | 66.3 (31.57) | 75.2 (24.85)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 36.9, 95% CI 2-sided [25.2 to 48.7]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5968, Mixed Models Analysis; LS Mean Difference = -3.2, 95% CI 2-sided [-14.9 to 8.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1471, Mixed Models Analysis; LS Mean Difference = 8.7, 95% CI 2-sided [-3.1 to 20.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1136, Mixed Models Analysis; LS Mean Difference = 9.5, 95% CI 2-sided [-2.3 to 21.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 22.4, 95% CI 2-sided [10.6 to 34.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1136, Mixed Models Analysis; LS Mean Difference = 9.5, 95% CI 2-sided [-2.3 to 21.3]

8. Secondary Outcome: Take Drug Again Effect at Hours 12, 24 and 36
Description: as for outcome 5
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm
  Hour 12 | 44.0 (20.63) | 54.7 (33.56) | 79.7 (22.37) | 45.8 (27.53) | 68.7 (30.31) | 78.9 (25.21)
  Hour 24 | 41.8 (21.79) | 55.5 (32.73) | 76.9 (26.77) | 41.0 (28.73) | 69.6 (28.34) | 78.3 (25.17)
  Hour 36 | 42.9 (20.40) | 53.9 (32.84) | 76.8 (25.12) | 41.1 (28.95) | 68.1 (31.99) | 76.8 (25.17)

9. Secondary Outcome: Overall Drug Liking: Peak Effect (Emax)
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking"). Emax = Maximum observed score.
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 50.8 (12.80) | 64.3 (24.00) | 80.8 (19.51) | 52.9 (21.33) | 74.0 (22.44) | 81.6 (23.15)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 28.5, 95% CI 2-sided [19.6 to 37.4]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6209, Mixed Models Analysis; LS Mean Difference = 2.2, 95% CI 2-sided [-6.7 to 11.1]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0997, Mixed Models Analysis; LS Mean Difference = 7.5, 95% CI 2-sided [-1.4 to 16.3]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 23.2, 95% CI 2-sided [14.4 to 32.1]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = 16.6, 95% CI 2-sided [7.7 to 25.5]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; LS Mean Difference = 13.3, 95% CI 2-sided [4.4 to 22.2]

10. Secondary Outcome: Overall Drug Liking: Mean Effect (Emean)
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking"). Emean = Average observed score.
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 50.19 (11.962) | 61.26 (24.489) | 75.70 (21.304) | 47.72 (20.715) | 69.94 (23.370) | 77.90 (23.077)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 29.9, 95% CI 2-sided [21.1 to 38.8]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5951, Mixed Models Analysis; LS Mean Difference = -2.4, 95% CI 2-sided [-11.2 to 6.4]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0841, Mixed Models Analysis; LS Mean Difference = 7.8, 95% CI 2-sided [-1.1 to 16.6]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.8, 95% CI 2-sided [11.0 to 28.6]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; LS Mean Difference = 14.5, 95% CI 2-sided [5.7 to 23.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0172, Mixed Models Analysis; LS Mean Difference = 10.8, 95% CI 2-sided [1.9 to 19.6]

11. Secondary Outcome: Overall Drug Liking: Minimum Effect (Emin)
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking"). Emin= Average observed score.
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 49.6 (11.40) | 58.5 (24.82) | 71.1 (25.28) | 43.6 (23.55) | 65.6 (25.87) | 74.3 (23.53)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 30.4, 95% CI 2-sided [21.0 to 39.9]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2166, Mixed Models Analysis; LS Mean Difference = -5.9, 95% CI 2-sided [-15.4 to 3.5]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0777, Mixed Models Analysis; LS Mean Difference = 8.5, 95% CI 2-sided [-1.0 to 18.0]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS Mean Difference = 16.0, 95% CI 2-sided [6.5 to 25.4]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0086, Mixed Models Analysis; LS Mean Difference = 12.7, 95% CI 2-sided [3.3 to 22.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0775, Mixed Models Analysis; LS Mean Difference = 8.5, 95% CI 2-sided [-0.9 to 18.0]

12. Secondary Outcome: Overall Drug Liking Effect at Hours 12, 24 and 36
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking").
Time Frame: 12, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm
  Hour 12 | 50.6 (12.78) | 61.2 (26.16) | 78.5 (20.86) | 51.8 (21.57) | 69.8 (23.19) | 78.1 (23.99)
  Hour 24 | 50.3 (11.84) | 62.7 (23.25) | 75.5 (24.26) | 44.8 (23.62) | 70.1 (24.53) | 78.1 (22.95)
  Hour 36 | 49.7 (11.41) | 59.9 (25.20) | 73.2 (25.03) | 46.6 (23.35) | 69.9 (25.43) | 77.6 (23.79)

13. Secondary Outcome: Any Drug Effects: Peak Effect (Emax)
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 8.8 (19.43) | 47.2 (38.45) | 82.4 (25.27) | 27.7 (35.77) | 56.0 (35.90) | 88.7 (20.52)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 61.2, 95% CI 2-sided [48.8 to 73.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis; LS Mean Difference = 18.8, 95% CI 2-sided [6.4 to 31.2]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 32.9, 95% CI 2-sided [20.5 to 45.3]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 47.2, 95% CI 2-sided [34.8 to 59.6]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 73.6, 95% CI 2-sided [61.1 to 86.0]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 38.4, 95% CI 2-sided [26.0 to 50.8]

14. Secondary Outcome: Any Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 1.105 (5.6058) | 20.129 (23.9971) | 40.199 (20.3489) | 4.539 (11.9639) | 26.566 (24.8693) | 48.328 (19.8494)
  AUE (0-2) | 3.090 (10.1113) | 57.504 (57.6543) | 112.910 (41.6661) | 10.734 (23.0043) | 69.059 (55.0442) | 124.617 (41.2197)
  AUE (0-8) | 5.949 (16.4695) | 140.152 (147.5551) | 283.770 (173.4241) | 53.242 (99.4186) | 167.137 (152.8249) | 354.391 (184.4799)
  AUE (0-12) | 5.949 (16.4695) | 156.652 (175.1035) | 317.270 (218.4262) | 107.180 (190.7655) | 176.199 (165.0887) | 392.828 (229.3565)
  AUE (0-24) | 13.762 (46.7425) | 157.059 (175.7028) | 345.301 (260.4659) | 218.805 (379.7129) | 184.137 (172.7494) | 402.516 (244.3471)
  AUE (0-36) | 23.324 (98.1331) | 157.059 (175.7028) | 345.488 (260.3746) | 235.117 (424.9088) | 186.387 (173.5877) | 402.703 (244.2750)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-1): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 43.9, 95% CI 2-sided [36.0 to 51.8]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.4154, Mixed Models Analysis; LS Mean Difference = 3.3, 95% CI 2-sided [-4.6 to 11.2]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 21.8, 95% CI 2-sided [13.9 to 29.7]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.4, 95% CI 2-sided [17.5 to 33.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 20.2, 95% CI 2-sided [12.3 to 28.1]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 18.9, 95% CI 2-sided [11.0 to 26.8]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-2): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 114.2, 95% CI 2-sided [97.1 to 131.3]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3985, Mixed Models Analysis; LS Mean Difference = 7.3, 95% CI 2-sided [-9.8 to 24.4]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 55.6, 95% CI 2-sided [38.5 to 72.8]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 65.9, 95% CI 2-sided [48.8 to 83.0]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 55.6, 95% CI 2-sided [38.5 to 72.7]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 54.1, 95% CI 2-sided [37.0 to 71.2]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-8): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 302.8, 95% CI 2-sided [248.8 to 356.8]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0824, Mixed Models Analysis; LS Mean Difference = 47.8, 95% CI 2-sided [-6.2 to 101.7]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 188.5, 95% CI 2-sided [134.6 to 242.5]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 162.0, 95% CI 2-sided [108.0 to 216.0]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 141.9, 95% CI 2-sided [87.9 to 195.8]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 135.7, 95% CI 2-sided [81.7 to 189.6]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-12): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 287.6, 95% CI 2-sided [219.1 to 356.1]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis; LS Mean Difference = 101.4, 95% CI 2-sided [32.9 to 169.8]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 218.5, 95% CI 2-sided [150.0 to 287.0]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 170.5, 95% CI 2-sided [102.0 to 239.0]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 158.6, 95% CI 2-sided [90.1 to 227.1]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 152.2, 95% CI 2-sided [83.7 to 220.7]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-24): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 185.9, 95% CI 2-sided [90.1 to 281.8]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 205.0, 95% CI 2-sided [109.2 to 300.8]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 221.0, 95% CI 2-sided [125.2 to 316.7]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 170.0, 95% CI 2-sided [74.1 to 265.8]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 185.7, 95% CI 2-sided [89.9 to 281.5]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0033, Mixed Models Analysis; LS Mean Difference = 144.9, 95% CI 2-sided [49.1 to 240.8]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; AUE (0-36): Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; LS Mean Difference = 170.0, 95% CI 2-sided [65.2 to 274.9]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = 211.4, 95% CI 2-sided [106.6 to 316.2]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 219.2, 95% CI 2-sided [114.5 to 324.0]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis; LS Mean Difference = 162.2, 95% CI 2-sided [57.3 to 267.0]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 185.9, 95% CI 2-sided [81.1 to 290.7]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; LS Mean Difference = 135.5, 95% CI 2-sided [30.7 to 240.4]

15. Secondary Outcome: Any Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.258 [0.25 to 24.02] | 1.017 [0.25 to 5.03] | 1.017 [0.27 to 4.00] | 0.758 [0.25 to 14.02] | 1.258 [0.25 to 8.03] | 1.017 [0.48 to 3.07]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.9, 95% CI 2-sided [-4.3 to -1.5]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = 2.8, 95% CI 2-sided [1.4 to 4.2]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7005, Mixed Models Analysis; LS Mean Difference = -0.3, 95% CI 2-sided [-1.7 to 1.1]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8440, Mixed Models Analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-1.3 to 1.5]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7295, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.6 to 1.1]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8757, Mixed Models Analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-1.3 to 1.5]

16. Secondary Outcome: Good Drug Effects: Peak Effect (Emax)
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 11.6 (24.91) | 48.1 (38.53) | 81.8 (24.54) | 24.2 (34.68) | 54.7 (36.16) | 84.3 (22.53)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 60.1, 95% CI 2-sided [47.4 to 72.9]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0514, Mixed Models Analysis; LS Mean Difference = 12.6, 95% CI 2-sided [-0.1 to 25.4]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 29.7, 95% CI 2-sided [17.0 to 42.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 43.0, 95% CI 2-sided [30.3 to 55.8]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 33.7, 95% CI 2-sided [21.0 to 46.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 36.4, 95% CI 2-sided [23.7 to 49.1]

17. Secondary Outcome: Good Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 0.805 (3.6598) | 20.727 (23.7958) | 40.992 (19.3835) | 5.254 (12.3129) | 28.234 (25.4785) | 44.656 (19.3060)
  AUE (0-2) | 3.055 (10.0140) | 56.352 (55.7819) | 110.430 (42.2789) | 10.543 (22.1051) | 71.305 (58.7340) | 114.953 (41.8081)
  AUE (0-8) | 9.063 (24.0659) | 130.758 (152.6257) | 261.813 (163.8714) | 40.418 (87.9945) | 159.750 (156.8189) | 332.352 (193.5146)
  AUE (0-12) | 9.250 (24.0378) | 148.195 (183.1627) | 282.875 (205.0344) | 77.855 (172.2503) | 168.688 (173.4909) | 372.414 (248.2861)
  AUE (0-24) | 17.469 (51.3009) | 148.883 (183.8413) | 297.656 (240.6821) | 161.043 (349.4292) | 180.875 (212.9759) | 380.414 (261.0990)
  AUE (0-36) | 26.844 (101.2648) | 148.883 (183.8413) | 297.844 (240.6209) | 171.355 (394.6735) | 180.875 (212.9759) | 380.602 (261.1626)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 39.5, 95% CI 2-sided [31.8 to 47.2]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.2739, Mixed Models Analysis; LS Mean Difference = 4.3, 95% CI 2-sided [-3.4 to 12.0]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 16.4, 95% CI 2-sided [8.7 to 24.1]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 27.4, 95% CI 2-sided [19.7 to 35.0]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 20.5, 95% CI 2-sided [12.8 to 28.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.7, 95% CI 2-sided [12.0 to 27.4]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 104.7, 95% CI 2-sided [87.7 to 121.8]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.4003, Mixed Models Analysis; LS Mean Difference = 7.3, 95% CI 2-sided [-9.8 to 24.3]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 43.6, 95% CI 2-sided [26.6 to 60.7]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 68.4, 95% CI 2-sided [51.3 to 85.4]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 54.3, 95% CI 2-sided [37.3 to 71.4]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 53.0, 95% CI 2-sided [36.0 to 70.1]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 292.5, 95% CI 2-sided [240.0 to 345.1]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2277, Mixed Models Analysis; LS Mean Difference = 32.2, 95% CI 2-sided [-20.3 to 84.7]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 173.1, 95% CI 2-sided [120.5 to 225.6]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 151.7, 95% CI 2-sided [99.1 to 204.2]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 129.8, 95% CI 2-sided [77.2 to 182.3]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 122.6, 95% CI 2-sided [70.0 to 175.1]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 295.3, 95% CI 2-sided [228.3 to 362.2]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0416, Mixed Models Analysis; LS Mean Difference = 69.6, 95% CI 2-sided [2.7 to 136.5]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 204.4, 95% CI 2-sided [137.5 to 271.3]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 160.5, 95% CI 2-sided [93.5 to 227.4]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = 133.0, 95% CI 2-sided [66.1 to 199.9]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 140.1, 95% CI 2-sided [73.1 to 207.0]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 219.5, 95% CI 2-sided [127.6 to 311.3]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; LS Mean Difference = 145.0, 95% CI 2-sided [53.2 to 236.8]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 200.2, 95% CI 2-sided [108.4 to 292.0]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; LS Mean Difference = 164.3, 95% CI 2-sided [72.4 to 256.1]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS Mean Difference = 146.6, 95% CI 2-sided [54.8 to 238.4]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis; LS Mean Difference = 132.7, 95% CI 2-sided [40.8 to 224.5]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 209.3, 95% CI 2-sided [108.3 to 310.3]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis; LS Mean Difference = 145.7, 95% CI 2-sided [44.7 to 246.6]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = 200.7, 95% CI 2-sided [99.7 to 301.6]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis; LS Mean Difference = 154.3, 95% CI 2-sided [53.3 to 255.3]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0046, Mixed Models Analysis; LS Mean Difference = 146.8, 95% CI 2-sided [45.9 to 247.8]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0171, Mixed Models Analysis; LS Mean Difference = 123.3, 95% CI 2-sided [22.3 to 224.3]

18. Secondary Outcome: Good Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.258 [0.25 to 24.02] | 1.017 [0.25 to 8.00] | 1.017 [0.27 to 4.00] | 0.517 [0.25 to 14.02] | 1.017 [0.25 to 8.03] | 1.017 [0.48 to 4.02]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; LS Mean Difference = -2.3, 95% CI 2-sided [-3.7 to -0.9]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0105, Mixed Models Analysis; LS Mean Difference = 1.9, 95% CI 2-sided [0.4 to 3.3]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7259, Mixed Models Analysis; LS Mean Difference = -0.3, 95% CI 2-sided [-1.7 to 1.2]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7813, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.6 to 1.2]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5235, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 1.0]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8512, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-1.6 to 1.3]

19. Secondary Outcome: Bad Drug Effects: Peak Effect (Emax)
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 5.8 (15.46) | 16.4 (26.76) | 26.5 (36.60) | 20.6 (35.67) | 16.9 (28.85) | 31.4 (32.67)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0883, Mixed Models Analysis; LS Mean Difference = 11.1, 95% CI 2-sided [-1.7 to 23.9]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0241, Mixed Models Analysis; LS Mean Difference = 14.8, 95% CI 2-sided [2.0 to 27.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0235, Mixed Models Analysis; LS Mean Difference = 14.8, 95% CI 2-sided [2.0 to 27.6]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0901, Mixed Models Analysis; LS Mean Difference = 11.1, 95% CI 2-sided [-1.7 to 23.9]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1313, Mixed Models Analysis; LS Mean Difference = 9.8, 95% CI 2-sided [-3.0 to 22.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0982, Mixed Models Analysis; LS Mean Difference = 10.8, 95% CI 2-sided [-2.0 to 23.6]

20. Secondary Outcome: Bad Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 0.652 (3.5995) | 0.977 (2.9225) | 4.359 (12.9297) | 0.445 (2.4294) | 0.918 (2.4707) | 3.621 (7.2682)
  AUE (0-2) | 1.270 (5.2494) | 8.164 (18.3516) | 16.023 (32.3331) | 2.359 (8.9454) | 4.840 (10.9280) | 17.059 (28.6213)
  AUE (0-8) | 2.527 (7.6234) | 28.984 (47.6235) | 60.133 (104.8279) | 22.195 (63.1674) | 38.191 (83.7177) | 81.777 (124.7723)
  AUE (0-12) | 2.527 (7.6234) | 29.984 (48.2808) | 71.195 (112.5641) | 41.570 (88.3012) | 46.691 (105.0132) | 96.715 (157.0901)
  AUE (0-24) | 10.340 (44.8420) | 30.203 (48.4810) | 85.477 (145.5365) | 138.039 (300.2416) | 50.348 (111.5406) | 102.434 (167.6105)
  AUE (0-36) | 19.715 (97.5206) | 30.578 (48.6353) | 85.852 (146.1250) | 169.352 (379.2034) | 51.473 (113.3471) | 102.621 (167.6904)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0351, Mixed Models Analysis; LS Mean Difference = 3.3, 95% CI 2-sided [0.2 to 6.3]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.8751, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-3.3 to 2.8]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0795, Mixed Models Analysis; LS Mean Difference = 2.7, 95% CI 2-sided [-0.3 to 5.8]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.8382, Mixed Models Analysis; LS Mean Difference = 0.3, 95% CI 2-sided [-2.7 to 3.4]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0289, Mixed Models Analysis; LS Mean Difference = 3.4, 95% CI 2-sided [0.4 to 6.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.7878, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-2.6 to 3.5]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS Mean Difference = 14.8, 95% CI 2-sided [5.6 to 24.0]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.821, Mixed Models Analysis; LS Mean Difference = 1.1, 95% CI 2-sided [-8.1 to 10.3]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis; LS Mean Difference = 12.3, 95% CI 2-sided [3.1 to 21.5]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.4454, Mixed Models Analysis; LS Mean Difference = 3.6, 95% CI 2-sided [-5.6 to 12.8]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0934, Mixed Models Analysis; LS Mean Difference = 7.9, 95% CI 2-sided [-1.3 to 17.1]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.1358, Mixed Models Analysis; LS Mean Difference = 7.0, 95% CI 2-sided [-2.2 to 16.2]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS Mean Difference = 59.8, 95% CI 2-sided [27.0 to 92.7]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2365, Mixed Models Analysis; LS Mean Difference = 19.7, 95% CI 2-sided [-13.1 to 52.6]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; LS Mean Difference = 43.9, 95% CI 2-sided [11.1 to 76.7]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0335, Mixed Models Analysis; LS Mean Difference = 35.7, 95% CI 2-sided [2.8 to 68.5]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0661, Mixed Models Analysis; LS Mean Difference = 30.8, 95% CI 2-sided [-2.1 to 63.6]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1074, Mixed Models Analysis; LS Mean Difference = 26.9, 95% CI 2-sided [-5.9 to 59.8]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; LS Mean Difference = 55.3, 95% CI 2-sided [15.8 to 94.9]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0543, Mixed Models Analysis; LS Mean Difference = 38.8, 95% CI 2-sided [-0.7 to 78.3]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis; LS Mean Difference = 50.2, 95% CI 2-sided [10.7 to 89.7]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0297, Mixed Models Analysis; LS Mean Difference = 43.9, 95% CI 2-sided [4.4 to 83.5]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0407, Mixed Models Analysis; LS Mean Difference = 41.3, 95% CI 2-sided [1.8 to 80.8]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.1710, Mixed Models Analysis; LS Mean Difference = 27.5, 95% CI 2-sided [-12.0 to 67.1]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.3362, Mixed Models Analysis; LS Mean Difference = -35.0, 95% CI 2-sided [-106.7 to 36.7]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 126.9, 95% CI 2-sided [55.2 to 198.5]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.1449, Mixed Models Analysis; LS Mean Difference = 53.2, 95% CI 2-sided [-18.5 to 124.8]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.2882, Mixed Models Analysis; LS Mean Difference = 38.7, 95% CI 2-sided [-33.0 to 110.4]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.1314, Mixed Models Analysis; LS Mean Difference = 55.0, 95% CI 2-sided [-16.6 to 126.7]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.5808, Mixed Models Analysis; LS Mean Difference = 20.1, 95% CI 2-sided [-51.6 to 91.8]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.1415, Mixed Models Analysis; LS Mean Difference = -66.2, 95% CI 2-sided [-154.6 to 22.3]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS Mean Difference = 149.1, 95% CI 2-sided [60.7 to 237.5]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.2423, Mixed Models Analysis; LS Mean Difference = 52.5, 95% CI 2-sided [-35.9 to 140.9]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.4980, Mixed Models Analysis; LS Mean Difference = 30.4, 95% CI 2-sided [-58.0 to 118.8]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.2253, Mixed Models Analysis; LS Mean Difference = 54.5, 95% CI 2-sided [-33.9 to 142.9]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.7945, Mixed Models Analysis; LS Mean Difference = 11.7, 95% CI 2-sided [-76.8 to 100.1]

21. Secondary Outcome: Bad Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.250 [0.25 to 24.02] | 0.267 [0.23 to 5.02] | 1.517 [0.25 to 24.02] | 0.308 [0.25 to 36.02] | 0.267 [0.25 to 12.02] | 1.758 [0.23 to 8.03]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; LS Mean Difference = -2.8, 95% CI 2-sided [-5.1 to -0.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = 4.2, 95% CI 2-sided [2.0 to 6.5]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5483, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-1.6 to 2.9]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5284, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-1.5 to 2.9]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1331, Mixed Models Analysis; LS Mean Difference = 1.7, 95% CI 2-sided [-0.5 to 3.9]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8732, Mixed Models Analysis; LS Mean Difference = 0.2, 95% CI 2-sided [-2.1 to 2.4]

22. Secondary Outcome: Feel Sick: Peak Effect (Emax)
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 3.1 (10.80) | 5.4 (15.14) | 8.8 (25.63) | 10.1 (26.35) | 2.6 (7.06) | 11.7 (28.16)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4555, Mixed Models Analysis; LS Mean Difference = 3.6, 95% CI 2-sided [-5.9 to 13.2]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1495, Mixed Models Analysis; LS Mean Difference = 6.9, 95% CI 2-sided [-2.5 to 16.4]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0200, Mixed Models Analysis; LS Mean Difference = 11.4, 95% CI 2-sided [1.8 to 20.9]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8668, Mixed Models Analysis; LS Mean Difference = -0.8, 95% CI 2-sided [-10.3 to 8.7]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3904, Mixed Models Analysis; LS Mean Difference = 4.1, 95% CI 2-sided [-5.3 to 13.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6524, Mixed Models Analysis; LS Mean Difference = 2.2, 95% CI 2-sided [-7.3 to 11.6]

23. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 0.539 (3.0494) | 0.629 (3.0605) | 0.957 (3.3182) | 0.035 (0.1463) | 0.039 (0.1435) | 0.996 (3.2217)
  AUE (0-2) | 0.727 (4.0198) | 3.004 (14.4372) | 4.160 (16.6354) | 1.051 (4.5067) | 0.758 (2.6560) | 2.762 (6.8438)
  AUE (0-8) | 0.984 (4.2307) | 5.176 (17.2686) | 13.387 (40.8525) | 12.324 (61.4559) | 5.281 (17.1483) | 15.449 (36.7603)
  AUE (0-12) | 0.984 (4.2307) | 5.176 (17.2686) | 13.387 (40.8525) | 12.949 (63.8914) | 6.156 (19.8004) | 19.137 (42.3860)
  AUE (0-24) | 8.797 (44.3081) | 5.645 (18.1099) | 13.387 (40.8525) | 64.699 (196.3450) | 7.406 (22.7994) | 19.605 (42.5054)
  AUE (0-36) | 18.359 (97.2004) | 6.582 (19.7796) | 13.387 (40.8525) | 83.449 (267.7102) | 7.594 (22.9559) | 21.855 (43.9416)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1771, Mixed Models Analysis; LS Mean Difference = 0.8, 95% CI 2-sided [-0.4 to 2.1]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3944, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1778, Mixed Models Analysis; LS Mean Difference = 0.8, 95% CI 2-sided [-0.4 to 2.1]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3960, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.6125, Mixed Models Analysis; LS Mean Difference = 0.3, 95% CI 2-sided [-0.9 to 1.5]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.9059, Mixed Models Analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-1.1 to 1.3]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.4585, Mixed Models Analysis; LS Mean Difference = 1.7, 95% CI 2-sided [-2.9 to 6.3]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.8986, Mixed Models Analysis; LS Mean Difference = 0.3, 95% CI 2-sided [-4.2 to 4.8]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3641, Mixed Models Analysis; LS Mean Difference = 2.1, 95% CI 2-sided [-2.5 to 6.7]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.9674, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-4.6 to 4.4]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.5744, Mixed Models Analysis; LS Mean Difference = 1.3, 95% CI 2-sided [-3.2 to 5.8]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3457, Mixed Models Analysis; LS Mean Difference = 2.2, 95% CI 2-sided [-2.4 to 6.7]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.6664, Mixed Models Analysis; LS Mean Difference = 3.7, 95% CI 2-sided [-13.3 to 20.8]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1949, Mixed Models Analysis; LS Mean Difference = 11.1, 95% CI 2-sided [-5.8 to 28.0]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2009, Mixed Models Analysis; LS Mean Difference = 11.1, 95% CI 2-sided [-6.0 to 28.1]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.6595, Mixed Models Analysis; LS Mean Difference = 3.8, 95% CI 2-sided [-13.1 to 20.7]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.3176, Mixed Models Analysis; LS Mean Difference = 8.6, 95% CI 2-sided [-8.3 to 25.5]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.6423, Mixed Models Analysis; LS Mean Difference = 4.0, 95% CI 2-sided [-12.9 to 20.9]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.4358, Mixed Models Analysis; LS Mean Difference = 6.8, 95% CI 2-sided [-10.5 to 24.2]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.1789, Mixed Models Analysis; LS Mean Difference = 11.7, 95% CI 2-sided [-5.4 to 28.9]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.1131, Mixed Models Analysis; LS Mean Difference = 14.0, 95% CI 2-sided [-3.3 to 31.3]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.5965, Mixed Models Analysis; LS Mean Difference = 4.6, 95% CI 2-sided [-12.6 to 21.8]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.3175, Mixed Models Analysis; LS Mean Difference = 8.7, 95% CI 2-sided [-8.5 to 25.9]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.6551, Mixed Models Analysis; LS Mean Difference = 3.9, 95% CI 2-sided [-13.3 to 21.0]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0354, Mixed Models Analysis; LS Mean Difference = -45.3, 95% CI 2-sided [-87.5 to -3.1]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0100, Mixed Models Analysis; LS Mean Difference = 55.2, 95% CI 2-sided [13.4 to 97.0]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.5379, Mixed Models Analysis; LS Mean Difference = 13.2, 95% CI 2-sided [-29.0 to 55.4]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.8768, Mixed Models Analysis; LS Mean Difference = -3.3, 95% CI 2-sided [-45.1 to 38.5]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.7031, Mixed Models Analysis; LS Mean Difference = 8.1, 95% CI 2-sided [-33.8 to 49.9]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.8507, Mixed Models Analysis; LS Mean Difference = -4, 95% CI 2-sided [-45.8 to 37.8]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0381, Mixed Models Analysis; LS Mean Difference = -62.3, 95% CI 2-sided [-121.2 to -3.5]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0318, Mixed Models Analysis; LS Mean Difference = 64.0, 95% CI 2-sided [5.7 to 122.3]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.6095, Mixed Models Analysis; LS Mean Difference = 15.2, 95% CI 2-sided [-43.6 to 74.1]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.6470, Mixed Models Analysis; LS Mean Difference = -13.6, 95% CI 2-sided [-71.9 to 44.8]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.8136, Mixed Models Analysis; LS Mean Difference = 7.0, 95% CI 2-sided [-51.4 to 65.4]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.6699, Mixed Models Analysis; LS Mean Difference = -12.6, 95% CI 2-sided [-71.0 to 45.7]

24. Secondary Outcome: Feel Sick: Time to Maximum (Peak) Effect (TEmax)
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.250 [0.25 to 36.00] | 0.267 [0.23 to 24.00] | 0.267 [0.25 to 3.03] | 0.267 [0.25 to 24.05] | 0.267 [0.25 to 12.02] | 0.267 [0.23 to 24.00]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1728, Mixed Models Analysis; LS Mean Difference = -1.6, 95% CI 2-sided [-3.9 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2616, Mixed Models Analysis; LS Mean Difference = 1.3, 95% CI 2-sided [-1.0 to 3.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7307, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-1.9 to 2.7]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5473, Mixed Models Analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-3.0 to 1.6]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4999, Mixed Models Analysis; LS Mean Difference = -0.8, 95% CI 2-sided [-3.1 to 1.5]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5592, Mixed Models Analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-3.0 to 1.6]

25. Secondary Outcome: Nausea: Peak Effect (Emax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 6.1 (18.90) | 11.5 (25.07) | 17.8 (32.11) | 9.5 (26.18) | 11.3 (23.47) | 22.0 (33.25)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0217, Mixed Models Analysis; LS Mean Difference = 13.3, 95% CI 2-sided [2.0 to 24.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5513, Mixed Models Analysis; LS Mean Difference = 3.4, 95% CI 2-sided [-7.8 to 14.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0469, Mixed Models Analysis; LS Mean Difference = 11.5, 95% CI 2-sided [0.2 to 22.8]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3604, Mixed Models Analysis; LS Mean Difference = 5.2, 95% CI 2-sided [-6.0 to 16.4]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2725, Mixed Models Analysis; LS Mean Difference = 6.2, 95% CI 2-sided [-5.0 to 17.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3461, Mixed Models Analysis; LS Mean Difference = 5.4, 95% CI 2-sided [-5.8 to 16.6]

26. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 1.551 (8.7270) | 1.313 (4.2183) | 3.867 (13.3986) | 0.043 (0.1510) | 0.281 (1.0395) | 2.797 (8.7018)
  AUE (0-2) | 3.309 (16.0847) | 6.938 (18.5123) | 11.500 (30.7880) | 0.520 (2.3602) | 3.813 (11.0316) | 9.398 (19.9006)
  AUE (0-8) | 5.801 (21.1576) | 17.656 (40.3906) | 34.102 (88.7640) | 12.465 (46.6764) | 15.453 (33.4096) | 39.648 (75.0136)
  AUE (0-12) | 5.801 (21.1576) | 17.656 (40.3906) | 40.602 (97.6330) | 16.340 (58.2244) | 18.828 (41.2148) | 41.523 (78.2852)
  AUE (0-24) | 13.613 (54.7055) | 17.656 (40.3906) | 52.508 (132.8214) | 76.402 (243.7336) | 21.203 (45.1793) | 42.992 (80.0147)
  AUE (0-36) | 22.988 (105.8442) | 17.844 (40.3199) | 52.508 (132.8214) | 94.777 (325.6554) | 21.391 (45.4013) | 43.742 (79.9894)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1828, Mixed Models Analysis; LS Mean Difference = 2.4, 95% CI 2-sided [-1.1 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3908, Mixed Models Analysis; LS Mean Difference = -1.5, 95% CI 2-sided [-5.0 to 1.9]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.2513, Mixed Models Analysis; LS Mean Difference = 2.0, 95% CI 2-sided [-1.5 to 5.5]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.5035, Mixed Models Analysis; LS Mean Difference = -1.2, 95% CI 2-sided [-4.6 to 2.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1452, Mixed Models Analysis; LS Mean Difference = 2.6, 95% CI 2-sided [-0.9 to 6.0]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.9303, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-3.6 to 3.3]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0283, Mixed Models Analysis; LS Mean Difference = 8.8, 95% CI 2-sided [0.9 to 16.7]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.4861, Mixed Models Analysis; LS Mean Difference = -2.7, 95% CI 2-sided [-10.5 to 5.0]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.1809, Mixed Models Analysis; LS Mean Difference = 5.3, 95% CI 2-sided [-2.5 to 13.2]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.8560, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-7.1 to 8.5]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.2385, Mixed Models Analysis; LS Mean Difference = 4.7, 95% CI 2-sided [-3.1 to 12.4]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3479, Mixed Models Analysis; LS Mean Difference = 3.7, 95% CI 2-sided [-4.1 to 11.5]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0185, Mixed Models Analysis; LS Mean Difference = 27.7, 95% CI 2-sided [4.7 to 50.6]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.5471, Mixed Models Analysis; LS Mean Difference = 6.9, 95% CI 2-sided [-15.8 to 29.7]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0367, Mixed Models Analysis; LS Mean Difference = 24.5, 95% CI 2-sided [1.5 to 47.4]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.3797, Mixed Models Analysis; LS Mean Difference = 10.1, 95% CI 2-sided [-12.6 to 32.9]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1557, Mixed Models Analysis; LS Mean Difference = 16.4, 95% CI 2-sided [-6.3 to 39.1]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2904, Mixed Models Analysis; LS Mean Difference = 12.2, 95% CI 2-sided [-10.5 to 34.9]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0467, Mixed Models Analysis; LS Mean Difference = 26.0, 95% CI 2-sided [0.4 to 51.6]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.4056, Mixed Models Analysis; LS Mean Difference = 10.7, 95% CI 2-sided [-14.6 to 36.0]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0738, Mixed Models Analysis; LS Mean Difference = 23.3, 95% CI 2-sided [-2.3 to 48.9]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.2987, Mixed Models Analysis; LS Mean Difference = 13.4, 95% CI 2-sided [-12.0 to 38.7]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0763, Mixed Models Analysis; LS Mean Difference = 22.9, 95% CI 2-sided [-2.4 to 48.2]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.3396, Mixed Models Analysis; LS Mean Difference = 12.3, 95% CI 2-sided [-13.1 to 37.6]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.2425, Mixed Models Analysis; LS Mean Difference = -33.2, 95% CI 2-sided [-89.1 to 22.7]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0281, Mixed Models Analysis; LS Mean Difference = 62.1, 95% CI 2-sided [6.8 to 117.5]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.4189, Mixed Models Analysis; LS Mean Difference = 22.9, 95% CI 2-sided [-33.0 to 78.8]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.8310, Mixed Models Analysis; LS Mean Difference = 6.0, 95% CI 2-sided [-49.4 to 61.4]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.2161, Mixed Models Analysis; LS Mean Difference = 34.8, 95% CI 2-sided [-20.6 to 90.1]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.8905, Mixed Models Analysis; LS Mean Difference = 3.9, 95% CI 2-sided [-51.5 to 59.2]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.1597, Mixed Models Analysis; LS Mean Difference = -51.8, 95% CI 2-sided [-124.2 to 20.6]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0525, Mixed Models Analysis; LS Mean Difference = 70.9, 95% CI 2-sided [-0.8 to 142.6]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.5294, Mixed Models Analysis; LS Mean Difference = 23.1, 95% CI 2-sided [-49.3 to 95.4]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.9126, Mixed Models Analysis; LS Mean Difference = -4.0, 95% CI 2-sided [-75.7 to 67.7]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.3418, Mixed Models Analysis; LS Mean Difference = 34.6, 95% CI 2-sided [-37.1 to 106.3]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.8833, Mixed Models Analysis; LS Mean Difference = -5.3, 95% CI 2-sided [-77.0 to 66.4]

27. Secondary Outcome: Nausea: Time to Maximum (Peak) Effect (TEmax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.250 [0.25 to 5.00] | 0.267 [0.25 to 36.00] | 0.267 [0.25 to 12.02] | 0.267 [0.25 to 36.02] | 0.267 [0.25 to 12.02] | 0.267 [0.23 to 6.00]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; LS Mean Difference = -3.6, 95% CI 2-sided [-6.1 to -1.2]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 4.3, 95% CI 2-sided [1.9 to 6.8]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8765, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-2.7 to 2.3]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4746, Mixed Models Analysis; LS Mean Difference = 0.9, 95% CI 2-sided [-1.6 to 3.3]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4607, Mixed Models Analysis; LS Mean Difference = -0.9, 95% CI 2-sided [-3.3 to 1.5]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2316, Mixed Models Analysis; LS Mean Difference = 1.5, 95% CI 2-sided [-1.0 to 3.9]

28. Secondary Outcome: Sleepy: Peak Effect (Emax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 24.7 (34.06) | 56.8 (35.54) | 72.0 (30.57) | 38.3 (38.32) | 59.2 (36.76) | 76.1 (25.88)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 38.8, 95% CI 2-sided [26.4 to 51.3]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0136, Mixed Models Analysis; LS Mean Difference = 15.8, 95% CI 2-sided [3.3 to 28.3]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; LS Mean Difference = 18.5, 95% CI 2-sided [6.1 to 31.0]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 36.1, 95% CI 2-sided [23.6 to 48.5]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0157, Mixed Models Analysis; LS Mean Difference = 15.4, 95% CI 2-sided [2.9 to 27.8]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 32.9, 95% CI 2-sided [20.5 to 45.3]

29. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 3.660 (11.1947) | 9.160 (12.4734) | 17.555 (18.6009) | 9.004 (18.9625) | 10.789 (17.0139) | 22.590 (19.7659)
  AUE (0-2) | 17.809 (35.0786) | 44.152 (38.4132) | 66.906 (46.9339) | 27.512 (43.9712) | 49.125 (49.5132) | 79.848 (46.1185)
  AUE (0-8) | 57.035 (117.1422) | 196.691 (178.5590) | 295.727 (204.5401) | 127.855 (188.5158) | 223.984 (196.8453) | 378.309 (195.1978)
  AUE (0-12) | 68.785 (151.3384) | 239.566 (244.9626) | 352.289 (260.5164) | 195.418 (271.9999) | 270.109 (253.5547) | 440.809 (232.3446)
  AUE (0-24) | 107.254 (299.1972) | 295.941 (314.6515) | 407.820 (342.4604) | 346.949 (494.5935) | 341.922 (407.7011) | 487.559 (284.8306)
  AUE (0-36) | 135.941 (402.8944) | 299.316 (316.1870) | 414.008 (349.3465) | 382.012 (585.0876) | 362.922 (486.0190) | 493.559 (290.1531)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 12.5, 95% CI 2-sided [6.4 to 18.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.2550, Mixed Models Analysis; LS Mean Difference = 3.5, 95% CI 2-sided [-2.6 to 9.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; LS Mean Difference = 10.4, 95% CI 2-sided [4.3 to 16.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0667, Mixed Models Analysis; LS Mean Difference = 5.7, 95% CI 2-sided [-0.4 to 11.8]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0075, Mixed Models Analysis; LS Mean Difference = 8.3, 95% CI 2-sided [2.3 to 14.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1354, Mixed Models Analysis; LS Mean Difference = 4.6, 95% CI 2-sided [-1.5 to 10.7]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 50.9, 95% CI 2-sided [34.2 to 67.5]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3905, Mixed Models Analysis; LS Mean Difference = 7.3, 95% CI 2-sided [-9.4 to 24.0]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; LS Mean Difference = 28.6, 95% CI 2-sided [11.9 to 45.3]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 29.6, 95% CI 2-sided [12.9 to 46.3]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis; LS Mean Difference = 22.9, 95% CI 2-sided [6.3 to 39.5]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; LS Mean Difference = 25.0, 95% CI 2-sided [8.4 to 41.6]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 248.4, 95% CI 2-sided [188.6 to 308.3]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0263, Mixed Models Analysis; LS Mean Difference = 68.2, 95% CI 2-sided [8.2 to 128.2]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 151.2, 95% CI 2-sided [91.3 to 211.1]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 165.4, 95% CI 2-sided [105.6 to 225.3]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; LS Mean Difference = 97.9, 95% CI 2-sided [38.3 to 157.6]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 138.4, 95% CI 2-sided [78.7 to 198.2]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 241.3, 95% CI 2-sided [162.8 to 319.9]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis; LS Mean Difference = 121.1, 95% CI 2-sided [42.4 to 199.9]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 164.4, 95% CI 2-sided [85.8 to 243.1]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 198.0, 95% CI 2-sided [119.4 to 276.6]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis; LS Mean Difference = 111.1, 95% CI 2-sided [32.8 to 189.4]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 168.1, 95% CI 2-sided [89.7 to 246.6]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0360, Mixed Models Analysis; LS Mean Difference = 128.4, 95% CI 2-sided [8.5 to 248.3]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS Mean Difference = 221.5, 95% CI 2-sided [101.2 to 341.7]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0388, Mixed Models Analysis; LS Mean Difference = 126.7, 95% CI 2-sided [6.6 to 246.8]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = 223.2, 95% CI 2-sided [103.2 to 343.2]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0787, Mixed Models Analysis; LS Mean Difference = 107.2, 95% CI 2-sided [-12.4 to 226.8]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0033, Mixed Models Analysis; LS Mean Difference = 181.3, 95% CI 2-sided [61.5 to 301.0]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.1688, Mixed Models Analysis; LS Mean Difference = 96.1, 95% CI 2-sided [-41.2 to 233.3]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS Mean Difference = 220.3, 95% CI 2-sided [82.6 to 358.0]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.1298, Mixed Models Analysis; LS Mean Difference = 106.0, 95% CI 2-sided [-31.5 to 243.5]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; LS Mean Difference = 210.4, 95% CI 2-sided [73.0 to 347.8]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.1189, Mixed Models Analysis; LS Mean Difference = 108.7, 95% CI 2-sided [-28.3 to 245.7]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0284, Mixed Models Analysis; LS Mean Difference = 153.6, 95% CI 2-sided [16.4 to 290.8]

30. Secondary Outcome: Sleepy: Time to Maximum (Peak) Effect (TEmax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm)to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.758 [0.25 to 24.02] | 2.025 [0.25 to 12.00] | 2.508 [0.25 to 12.02] | 2.000 [0.25 to 14.03] | 2.017 [0.27 to 12.02] | 2.033 [0.52 to 6.02]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0327, Mixed Models Analysis; LS Mean Difference = -1.8, 95% CI 2-sided [-3.4 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS Mean Difference = 2.6, 95% CI 2-sided [1.0 to 4.2]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7508, Mixed Models Analysis; LS Mean Difference = -0.3, 95% CI 2-sided [-1.9 to 1.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1868, Mixed Models Analysis; LS Mean Difference = 1.1, 95% CI 2-sided [-0.5 to 2.7]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9944, Mixed Models Analysis; LS Mean Difference = 0.0, 95% CI 2-sided [-1.6 to 1.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2322, Mixed Models Analysis; LS Mean Difference = 1.0, 95% CI 2-sided [-0.6 to 2.6]

31. Secondary Outcome: Dizzy: Peak Effect (Emax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | 3.6 (12.27) | 23.4 (32.63) | 30.6 (36.58) | 12.0 (28.21) | 19.5 (31.56) | 39.3 (37.92)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 28.2, 95% CI 2-sided [16.8 to 39.6]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1421, Mixed Models Analysis; LS Mean Difference = 8.4, 95% CI 2-sided [-2.8 to 19.6]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS Mean Difference = 20.9, 95% CI 2-sided [9.5 to 32.2]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; LS Mean Difference = 15.8, 95% CI 2-sided [4.5 to 27.0]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1974, Mixed Models Analysis; LS Mean Difference = 7.4, 95% CI 2-sided [-3.9 to 18.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = 19.5, 95% CI 2-sided [8.3 to 30.8]

32. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 0.125 (0.5425) | 7.117 (15.3098) | 10.117 (15.9090) | 1.238 (4.8747) | 6.207 (12.4631) | 14.043 (17.1328)
  AUE (0-2) | 0.922 (3.0851) | 24.008 (41.3549) | 28.758 (39.5123) | 2.738 (10.8592) | 18.402 (33.2777) | 35.691 (44.1487)
  AUE (0-8) | 1.844 (6.2523) | 47.297 (82.8121) | 75.828 (117.4212) | 23.934 (82.1109) | 41.410 (79.0200) | 117.738 (146.9677)
  AUE (0-12) | 1.906 (6.2536) | 48.422 (85.1544) | 83.266 (131.6787) | 47.684 (145.0991) | 42.160 (79.5674) | 122.551 (150.8804)
  AUE (0-24) | 10.094 (49.8279) | 49.922 (88.2865) | 85.484 (136.4813) | 120.934 (324.0852) | 43.754 (81.6192) | 122.895 (150.6660)
  AUE (0-36) | 19.844 (102.7158) | 50.109 (88.1834) | 85.859 (136.2835) | 135.559 (386.0688) | 44.129 (81.4783) | 123.457 (150.3432)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 12.2, 95% CI 2-sided [7.1 to 17.4]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.6868, Mixed Models Analysis; LS Mean Difference = 1.0, 95% CI 2-sided [-4.1 to 6.2]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis; LS Mean Difference = 7.3, 95% CI 2-sided [2.2 to 12.5]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0229, Mixed Models Analysis; LS Mean Difference = 5.9, 95% CI 2-sided [0.8 to 11.1]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.2168, Mixed Models Analysis; LS Mean Difference = 3.2, 95% CI 2-sided [-1.9 to 8.3]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0096, Mixed Models Analysis; LS Mean Difference = 6.8, 95% CI 2-sided [1.7 to 11.9]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 33.0, 95% CI 2-sided [20.0 to 45.9]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.8009, Mixed Models Analysis; LS Mean Difference = 1.6, 95% CI 2-sided [-11.2 to 14.4]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0086, Mixed Models Analysis; LS Mean Difference = 17.4, 95% CI 2-sided [4.5 to 30.3]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis; LS Mean Difference = 17.2, 95% CI 2-sided [4.4 to 30.0]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.4224, Mixed Models Analysis; LS Mean Difference = 5.2, 95% CI 2-sided [-7.6 to 18.0]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 22.6, 95% CI 2-sided [9.8 to 35.5]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 96.1, 95% CI 2-sided [57.9 to 134.2]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2530, Mixed Models Analysis; LS Mean Difference = 21.9, 95% CI 2-sided [-15.8 to 59.7]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 78.6, 95% CI 2-sided [40.5 to 116.8]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0414, Mixed Models Analysis; LS Mean Difference = 39.3, 95% CI 2-sided [1.6 to 77.1]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1329, Mixed Models Analysis; LS Mean Difference = 28.9, 95% CI 2-sided [-8.9 to 66.6]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0187, Mixed Models Analysis; LS Mean Difference = 45.5, 95% CI 2-sided [7.7 to 83.2]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; LS Mean Difference = 76.9, 95% CI 2-sided [31.9 to 121.9]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0456, Mixed Models Analysis; LS Mean Difference = 45.4, 95% CI 2-sided [0.9 to 89.9]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS Mean Difference = 82.8, 95% CI 2-sided [37.8 to 127.7]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0812, Mixed Models Analysis; LS Mean Difference = 39.6, 95% CI 2-sided [-5.0 to 84.1]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.1174, Mixed Models Analysis; LS Mean Difference = 35.5, 95% CI 2-sided [-9.0 to 80.0]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0427, Mixed Models Analysis; LS Mean Difference = 46.1, 95% CI 2-sided [1.5 to 90.6]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.9318, Mixed Models Analysis; LS Mean Difference = 3.0, 95% CI 2-sided [-66.9 to 73.0]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; LS Mean Difference = 110.4, 95% CI 2-sided [41.2 to 179.6]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0226, Mixed Models Analysis; LS Mean Difference = 81.5, 95% CI 2-sided [11.6 to 151.4]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.3629, Mixed Models Analysis; LS Mean Difference = 32.0, 95% CI 2-sided [-37.3 to 101.2]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.3077, Mixed Models Analysis; LS Mean Difference = 35.9, 95% CI 2-sided [-33.4 to 105.1]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.2662, Mixed Models Analysis; LS Mean Difference = 39.1, 95% CI 2-sided [-30.1 to 108.4]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.7875, Mixed Models Analysis; LS Mean Difference = -11.4, 95% CI 2-sided [-94.7 to 71.9]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0066, Mixed Models Analysis; LS Mean Difference = 115.0, 95% CI 2-sided [32.6 to 197.4]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0540, Mixed Models Analysis; LS Mean Difference = 81.7, 95% CI 2-sided [-1.4 to 164.9]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.6014, Mixed Models Analysis; LS Mean Difference = 21.8, 95% CI 2-sided [-60.6 to 104.3]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.3885, Mixed Models Analysis; LS Mean Difference = 36.1, 95% CI 2-sided [-46.3 to 118.5]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.4801, Mixed Models Analysis; LS Mean Difference = 29.5, 95% CI 2-sided [-52.9 to 112.0]

33. Secondary Outcome: Dizzy: Time to Maximum (Peak) Effect (TEmax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.250 [0.25 to 8.00] | 0.758 [0.25 to 36.02] | 0.767 [0.25 to 24.02] | 0.258 [0.25 to 14.02] | 0.292 [0.25 to 13.98] | 0.758 [0.23 to 8.03]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5494, Mixed Models Analysis; LS Mean Difference = -0.6, 95% CI 2-sided [-2.5 to 1.4]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0626, Mixed Models Analysis; LS Mean Difference = 1.8, 95% CI 2-sided [-0.1 to 3.8]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7216, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-1.6 to 2.3]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3647, Mixed Models Analysis; LS Mean Difference = 0.9, 95% CI 2-sided [-1.0 to 2.8]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4456, Mixed Models Analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-2.7 to 1.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0500, Mixed Models Analysis; LS Mean Difference = 1.9, 95% CI 2-sided [0.0 to 3.9]

34. Secondary Outcome: Pupillometry: Peak Effect (Emax)
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. Emax = Maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
mm | -0.8 (0.38) | -2.0 (0.71) | -2.7 (0.72) | -2.4 (0.71) | -2.1 (0.63) | -3.0 (0.76)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.51, 95% CI 2-sided [-0.69 to -0.34]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.69, 95% CI 2-sided [-1.86 to -1.52]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.80, 95% CI 2-sided [-0.97 to -0.63]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.40, 95% CI 2-sided [-1.58 to -1.23]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.74, 95% CI 2-sided [-0.91 to -0.56]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.29, 95% CI 2-sided [-1.46 to -1.11]

35. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 5.160 (0.7979) | 4.022 (0.7658) | 3.599 (0.6554) | 5.039 (0.7893) | 3.986 (0.6847) | 3.489 (0.6738)
  AUE (0-2) | 10.164 (1.5890) | 7.564 (1.3695) | 6.226 (1.0741) | 9.889 (1.6078) | 7.384 (1.2278) | 5.927 (1.0310)
  AUE (0-8) | 41.088 (6.4135) | 30.129 (5.7346) | 23.795 (4.0637) | 33.605 (6.4972) | 29.298 (5.4769) | 21.913 (3.6297)
  AUE (0-12) | 62.550 (9.6352) | 47.586 (9.5615) | 38.713 (7.6202) | 46.155 (8.8631) | 46.136 (8.9456) | 35.088 (6.4060)
  AUE (0-24) | 125.791 (19.2063) | 103.711 (19.5429) | 91.216 (17.4729) | 83.530 (14.6930) | 102.183 (17.7741) | 83.832 (17.6410)
  AUE (0-36) | 188.828 (29.4183) | 162.961 (29.2071) | 149.454 (25.4599) | 130.199 (23.0719) | 161.977 (26.8529) | 141.638 (28.1687)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.59, 95% CI 2-sided [-1.75 to -1.42]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3309, Mixed Models Analysis; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.58, 95% CI 2-sided [-0.74 to -0.42]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.09, 95% CI 2-sided [-1.25 to -0.92]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.42, 95% CI 2-sided [-0.59 to -0.26]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.04, 95% CI 2-sided [-1.21 to -0.88]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.03, 95% CI 2-sided [-4.37 to -3.69]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.2475, Mixed Models Analysis; LS Mean Difference = -0.20, 95% CI 2-sided [-0.54 to 0.14]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.61, 95% CI 2-sided [-1.96 to -1.27]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.62, 95% CI 2-sided [-2.96 to -2.27]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.34, 95% CI 2-sided [-1.68 to -1.00]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.42, 95% CI 2-sided [-2.76 to -2.08]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.91, 95% CI 2-sided [-13.21 to -10.60]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -7.23, 95% CI 2-sided [-8.54 to -5.93]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -7.90, 95% CI 2-sided [-9.20 to -6.59]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.24, 95% CI 2-sided [-12.55 to -9.94]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -6.35, 95% CI 2-sided [-7.65 to -5.05]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.36, 95% CI 2-sided [-11.67 to -9.05]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.37, 95% CI 2-sided [-13.16 to -9.58]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -16.07, 95% CI 2-sided [-17.86 to -14.28]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.73, 95% CI 2-sided [-13.53 to -9.93]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -15.71, 95% CI 2-sided [-17.51 to -13.91]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.88, 95% CI 2-sided [-10.67 to -7.09]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -14.19, 95% CI 2-sided [-15.99 to -12.39]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.8784, Mixed Models Analysis; LS Mean Difference = -0.26, 95% CI 2-sided [-3.63 to 3.11]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -41.66, 95% CI 2-sided [-45.02 to -38.29]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -19.63, 95% CI 2-sided [-23.01 to -16.25]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -22.28, 95% CI 2-sided [-25.67 to -18.90]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.50, 95% CI 2-sided [-15.86 to -9.14]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -20.59, 95% CI 2-sided [-23.98 to -17.21]
Statistical Analysis 31: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 10.64, 95% CI 2-sided [5.75 to 15.54]
Statistical Analysis 32: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -57.74, 95% CI 2-sided [-62.63 to -52.85]
Statistical Analysis 33: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -22.18, 95% CI 2-sided [-27.09 to -17.27]
Statistical Analysis 34: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -24.91, 95% CI 2-sided [-29.83 to -20.00]
Statistical Analysis 35: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.53, 95% CI 2-sided [-18.41 to -8.64]
Statistical Analysis 36: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -23.70, 95% CI 2-sided [-28.62 to -18.78]

36. Secondary Outcome: Pupillometry: Time to Maximum (Peak) Effect (TEmax)
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 2.275 [0.52 to 36.02] | 1.517 [0.52 to 6.02] | 1.517 [0.53 to 5.02] | 12.050 [5.00 to 14.03] | 1.775 [0.52 to 5.02] | 1.533 [0.50 to 6.02]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.73, 95% CI 2-sided [-11.90 to -7.57]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 5.16, 95% CI 2-sided [2.99 to 7.32]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9766, Mixed Models Analysis; LS Mean Difference = 0.03, 95% CI 2-sided [-2.13 to 2.20]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.61, 95% CI 2-sided [-6.78 to -2.44]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7242, Mixed Models Analysis; LS Mean Difference = -0.39, 95% CI 2-sided [-2.55 to 1.78]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.45, 95% CI 2-sided [-6.62 to -2.28]

37. Other Pre Specified Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-1 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time 0 to x hours (0-x).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 50.020 (2.7443) | 57.770 (11.2102) | 64.820 (14.3058) | 50.703 (3.2294) | 61.125 (12.7119) | 69.734 (12.6273)
  AUE (0-8) | 399.957 (8.2973) | 431.973 (80.0157) | 492.578 (112.1774) | 404.578 (71.1457) | 465.945 (110.9382) | 531.586 (110.7145)
  AUE (0-12) | 600.645 (8.1980) | 640.223 (111.0897) | 704.328 (140.9602) | 616.203 (130.7196) | 677.320 (147.0075) | 758.336 (160.5459)
  AUE (0-24) | 1202.863 (9.1566) | 1267.410 (197.1640) | 1337.016 (241.1654) | 1203.828 (289.3240) | 1285.289 (209.4193) | 1398.836 (237.2094)
  AUE (0-36) | 1805.113 (11.7017) | 1893.848 (298.9190) | 1955.953 (326.5777) | 1783.578 (361.8779) | 1907.414 (310.0402) | 2024.711 (347.2035)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.0, 95% CI 2-sided [14.6 to 23.5]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.8048, Mixed Models Analysis; LS Mean Difference = 0.6, 95% CI 2-sided [-3.9 to 5.0]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 8.6, 95% CI 2-sided [4.2 to 13.1]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 11.0, 95% CI 2-sided [6.5 to 15.4]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS Mean Difference = 7.1, 95% CI 2-sided [2.7 to 11.6]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; LS Mean Difference = 7.6, 95% CI 2-sided [3.2 to 12.1]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 127.4, 95% CI 2-sided [93.6 to 161.2]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.7837, Mixed Models Analysis; LS Mean Difference = 4.7, 95% CI 2-sided [-29.1 to 38.5]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 65.8, 95% CI 2-sided [32.0 to 99.6]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 66.3, 95% CI 2-sided [32.5 to 100.1]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 60.3, 95% CI 2-sided [26.5 to 94.1]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.0640, Mixed Models Analysis; LS Mean Difference = 31.9, 95% CI 2-sided [-1.9 to 65.7]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 142.6, 95% CI 2-sided [94.5 to 190.7]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.5169, Mixed Models Analysis; LS Mean Difference = 15.8, 95% CI 2-sided [-32.3 to 63.9]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS Mean Difference = 81.3, 95% CI 2-sided [33.2 to 129.3]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; LS Mean Difference = 77.1, 95% CI 2-sided [29.1 to 125.2]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0098, Mixed Models Analysis; LS Mean Difference = 63.6, 95% CI 2-sided [15.6 to 111.7]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.1078, Mixed Models Analysis; LS Mean Difference = 39.4, 95% CI 2-sided [-8.7 to 87.4]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 196.0, 95% CI 2-sided [116.9 to 275.1]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.9726, Mixed Models Analysis; LS Mean Difference = 1.4, 95% CI 2-sided [-77.7 to 80.5]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis; LS Mean Difference = 114.1, 95% CI 2-sided [35.0 to 193.2]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0392, Mixed Models Analysis; LS Mean Difference = 83.3, 95% CI 2-sided [4.2 to 162.4]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0883, Mixed Models Analysis; LS Mean Difference = 68.7, 95% CI 2-sided [-10.4 to 147.8]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.1100, Mixed Models Analysis; LS Mean Difference = 64.4, 95% CI 2-sided [-14.7 to 143.5]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 242.9, 95% CI 2-sided [138.6 to 347.2]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.6906, Mixed Models Analysis; LS Mean Difference = -21.0, 95% CI 2-sided [-125.3 to 83.2]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0259, Mixed Models Analysis; LS Mean Difference = 118.7, 95% CI 2-sided [14.5 to 223.0]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0525, Mixed Models Analysis; LS Mean Difference = 103.2, 95% CI 2-sided [-1.1 to 207.5]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.2558, Mixed Models Analysis; LS Mean Difference = 60.2, 95% CI 2-sided [-44.1 to 164.4]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0952, Mixed Models Analysis; LS Mean Difference = 88.6, 95% CI 2-sided [-15.7 to 192.9]

38. Other Pre Specified Outcome: Drug Liking: Time to Maximum (Peak) Effect (TEmax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.267 [0.25 to 5.02] | 1.017 [0.25 to 24.02] | 1.017 [0.27 to 14.02] | 0.758 [0.25 to 14.02] | 1.017 [0.25 to 24.02] | 1.008 [0.25 to 24.02]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0298, Mixed Models Analysis; LS Mean Difference = -1.8, 95% CI 2-sided [-3.3 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = 2.7, 95% CI 2-sided [1.1 to 4.3]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6450, Mixed Models Analysis; LS Mean Difference = -0.4, 95% CI 2-sided [-2.0 to 1.2]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0962, Mixed Models Analysis; LS Mean Difference = 1.3, 95% CI 2-sided [-0.2 to 2.9]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1930, Mixed Models Analysis; LS Mean Difference = -1.0, 95% CI 2-sided [-2.6 to 0.5]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0310, Mixed Models Analysis; LS Mean Difference = 1.7, 95% CI 2-sided [0.2 to 3.3]

39. Other Pre Specified Outcome: High: Area Under Effect Curve (AUE) From 0-1 Hour, 0-8 Hour, 0-12 Hour, 0-24 Hour and 0-36 Hour
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time 0 to x hours (0-x).
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours*mm
  AUE (0-1) | 0.785 (4.1738) | 20.203 (22.8004) | 40.801 (20.3235) | 4.473 (11.7536) | 27.465 (24.2206) | 45.836 (20.4802)
  AUE (0-8) | 6.512 (16.7072) | 119.055 (142.3080) | 257.527 (163.9543) | 39.145 (85.5494) | 153.941 (150.3297) | 322.250 (187.7896)
  AUE (0-12) | 6.512 (16.7072) | 131.805 (168.5472) | 277.715 (201.6860) | 78.582 (166.6578) | 160.004 (160.4458) | 355.250 (237.6863)
  AUE (0-24) | 24.199 (69.6362) | 131.930 (168.8668) | 282.902 (215.7112) | 161.613 (319.3473) | 171.129 (180.2282) | 362.531 (252.5074)
  AUE (0-36) | 34.137 (110.6283) | 132.305 (170.0009) | 282.902 (215.7112) | 168.176 (337.3448) | 173.379 (181.7041) | 362.531 (252.5074)
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 41.5, 95% CI 2-sided [33.9 to 49.0]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3763, Mixed Models Analysis; LS Mean Difference = 3.4, 95% CI 2-sided [-4.2 to 10.9]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 18.3, 95% CI 2-sided [10.7 to 25.8]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.6, 95% CI 2-sided [19.1 to 34.1]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 20.7, 95% CI 2-sided [13.1 to 28.2]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.3, 95% CI 2-sided [11.8 to 26.8]
Statistical Analysis 7: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 284.3, 95% CI 2-sided [232.9 to 335.8]
Statistical Analysis 8: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.2336, Mixed Models Analysis; LS Mean Difference = 31.2, 95% CI 2-sided [-20.4 to 82.8]
Statistical Analysis 9: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 167.3, 95% CI 2-sided [115.7 to 218.9]
Statistical Analysis 10: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 148.3, 95% CI 2-sided [96.8 to 199.7]
Statistical Analysis 11: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 135.6, 95% CI 2-sided [84.0 to 187.2]
Statistical Analysis 12: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 113.6, 95% CI 2-sided [62.1 to 165.0]
Statistical Analysis 13: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 278.3, 95% CI 2-sided [213.2 to 343.3]
Statistical Analysis 14: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0322, Mixed Models Analysis; LS Mean Difference = 71.3, 95% CI 2-sided [6.1 to 136.5]
Statistical Analysis 15: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 195.4, 95% CI 2-sided [130.2 to 260.5]
Statistical Analysis 16: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 154.3, 95% CI 2-sided [89.2 to 219.3]
Statistical Analysis 17: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 143.2, 95% CI 2-sided [78.0 to 208.4]
Statistical Analysis 18: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 126.7, 95% CI 2-sided [61.7 to 191.8]
Statistical Analysis 19: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 202.4, 95% CI 2-sided [118.4 to 286.4]
Statistical Analysis 20: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; LS Mean Difference = 137.6, 95% CI 2-sided [53.3 to 221.8]
Statistical Analysis 21: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 192.9, 95% CI 2-sided [108.7 to 277.2]
Statistical Analysis 22: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; LS Mean Difference = 147.0, 95% CI 2-sided [63.0 to 231.1]
Statistical Analysis 23: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; LS Mean Difference = 148.1, 95% CI 2-sided [63.9 to 232.4]
Statistical Analysis 24: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.0110, Mixed Models Analysis; LS Mean Difference = 109.6, 95% CI 2-sided [25.5 to 193.6]
Statistical Analysis 25: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 196.0, 95% CI 2-sided [107.4 to 284.6]
Statistical Analysis 26: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; LS Mean Difference = 133.9, 95% CI 2-sided [45.0 to 222.8]
Statistical Analysis 27: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 190.9, 95% CI 2-sided [102.1 to 279.8]
Statistical Analysis 28: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; LS Mean Difference = 138.9, 95% CI 2-sided [50.3 to 227.6]
Statistical Analysis 29: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; LS Mean Difference = 147.8, 95% CI 2-sided [59.0 to 236.7]
Statistical Analysis 30: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.0273, Mixed Models Analysis; LS Mean Difference = 100.0, 95% CI 2-sided [11.3 to 188.6]

40. Other Pre Specified Outcome: High: Time to Maximum (Peak) Effect (TEmax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
hours | 0.250 [0.25 to 24.02] | 1.017 [0.25 to 6.00] | 1.017 [0.27 to 4.00] | 0.767 [0.25 to 14.03] | 1.017 [0.25 to 8.03] | 1.017 [0.48 to 3.03]
Statistical Analysis 1: Comparison: ALO-02 60 Mg-I vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -3.4, 95% CI 2-sided [-5.0 to -1.8]
Statistical Analysis 2: Comparison: Placebo vs ALO-02 60 Mg-I; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS Mean Difference = 2.9, 95% CI 2-sided [1.3 to 4.4]
Statistical Analysis 3: Comparison: ALO-02 60 mg- C vs OXY 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8478, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.7 to 1.4]
Statistical Analysis 4: Comparison: Placebo vs ALO-02 60 mg- C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6192, Mixed Models Analysis; LS Mean Difference = -0.4, 95% CI 2-sided [-1.9 to 1.2]
Statistical Analysis 5: Comparison: ALO-02 40 Mg-C vs OXY 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8857, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-1.7 to 1.4]
Statistical Analysis 6: Comparison: Placebo vs ALO-02 40 Mg-C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5092, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-2.1 to 1.0]

41. Other Pre Specified Outcome: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of Oxycodone, Oxymorphone and Noroxycodone
Description: Cmax[dn]=Dose normalized maximum observed plasma concentration of participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the Pharmacokinetic (PK) parameters of interest. Here 'n' signifies those participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter/milligram
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 38 | 37 | 36
nanogram/milliliter/milligram
  Oxycodone (n= 36, 37, 38, 37, 36) | 1.989 (0.62042) | 1.672 (0.40716) | 0.4978 (0.15863) | 1.923 (0.54296) | 1.514 (0.42099)
  Oxymorphone (n= 36, 36, 38, 37, 35) | 0.03271 (0.0155) | 0.02847 (0.0149) | 0.0068 (0.00365) | 0.03182 (0.0161) | 0.02419 (0.0118)
  Noroxycodone (n= 36, 37, 38, 37, 36) | 1.295 (0.37231) | 1.123 (0.29543) | 0.3672 (0.18111) | 1.343 (0.36175) | 1.026 (0.33231)

42. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Naltrexone and 6-beta-naltrexol
Description: Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- ALO-02 40 Mg-C: Single dose of ALO-02 40mg/4.8 mg crushed tablet (ALO-02 40 mg-C) solution orally in either of the first to sixth intervention periods.
- ALO-02 60 Mg-C: Single dose of ALO-02 60 mg/7.2 mg crushed tablet (ALO-02 60 mg-C) solution orally in either of the first to sixth intervention periods.
Arm/Group | ALO-02 40 Mg-C | ALO-02 60 Mg-I | ALO-02 60 Mg-C
Number analyzed (Participants) | 36 | 38 | 37
nanogram per milliliter (ng/mL)
  Naltrexone | 1.389 (1.4633) | 0.01808 (0.11145) | 2.331 (2.4498)
  6-beta-naltrexol | 8.516 (2.4847) | 0.3012 (1.8325) | 13.70 (3.1369)

43. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Oxycodone, Oxymorphone and Noroxycodone
Description: Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest. Here 'n' signifies those participants who were evaluable for specified category.
Measure: Median (Full Range); unit: hours
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 38 | 37 | 36
hours
  Oxycodone (n= 36, 37, 38, 37, 36) | 1.03 [0.533 to 2.55] | 1.03 [0.283 to 3.07] | 12.1 [3.03 to 14.1] | 0.583 [0.533 to 1.55] | 1.04 [0.300 to 2.55]
  Oxymorphone (n= 36, 36, 37, 37, 35) | 0.559 [0.300 to 1.58] | 0.567 [0.283 to 3.07] | 14.0 [8.07 to 24.1] | 0.567 [0.300 to 1.07] | 0.550 [0.300 to 2.55]
  Noroxycodone (n= 36, 37, 38, 37, 36) | 1.03 [0.533 to 3.03] | 1.07 [0.533 to 3.07] | 14.1 [3.03 to 24.1] | 0.600 [0.533 to 3.08] | 1.05 [0.300 to 5.03]

44. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Naltrexone and 6-beta-naltrexol
Description: Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 43
Measure: Median (Full Range); unit: hour
Arm/Group | ALO-02 40 Mg-C | ALO-02 60 Mg-I | ALO-02 60 Mg-C
Number analyzed (Participants) | 36 | 38 | 37
hour
  Naltrexone (n= 36, 1, 37) | 0.550 [0.283 to 1.58] | 1.58 [1.58 to 1.58] | 0.550 [0.283 to 1.07]
  6-beta-naltrexol (n= 36, 19, 37) | 0.567 [0.367 to 2.55] | 1.55 [0.000 to 36.1] | 0.550 [0.283 to 1.55]

45. Other Pre Specified Outcome: Plasma Terminal Half-Life (t1/2) of Oxycodone
Description: Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Median (Full Range); unit: hours
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 35 | 37 | 36
hours | 4.470 [3.14 to 5.82] | 4.240 [3.07 to 5.91] | 9.340 [5.67 to 12.4] | 4.300 [3.02 to 5.81] | 4.195 [3.20 to 5.35]

46. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUC) From 0-1 Hour, 0-2 Hour, 0-8 Hour 0-12 Hour and 0-24 Hour of Oxycodone
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Participants who received oxycodone were reported.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 38 | 37 | 36
nanogram*hour/milliliter (ng*hr/mL)
  AUC (0-1) | 45.21 (19.256) | 37.60 (13.292) | 0.02102 (0.05715) | 72.25 (24.141) | 53.38 (19.223)
  AUC (0-2) | 103.5 (29.463) | 88.12 (20.159) | 0.7834 (0.42296) | 157.5 (37.317) | 120.0 (34.767)
  AUC (0-8) | 276.8 (72.686) | 265.0 (55.929) | 79.08 (19.900) | 405.5 (98.993) | 366.5 (88.598)
  AUC (0-12) | 319.6 (87.905) | 314.1 (72.753) | 181.6 (43.706) | 464.8 (121.19) | 451.5 (116.62)
  AUC (0-24) | 356.2 (104.68) | 355.9 (91.851) | 455.3 (118.50) | 513.9 (143.01) | 527.8 (149.84)

47. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Oxycodone
Description: Area under the plasma concentration time-curve from zero to the last quantifiable concentration (AUClast). Participants who received oxycodone were reported.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 38 | 37 | 36
ng*hr/mL | 361.6 (108.39) | 361.6 (95.617) | 575.8 (150.15) | 521.0 (147.32) | 538.6 (155.71)

48. Other Pre Specified Outcome: Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)dn] of Oxycodone
Description: [AUC (0 - ∞)dn]= Dose normalized area under the plasma concentration versus time curve [AUC(dn)] from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0- t) plus AUC (t - ∞). Participants who received oxycodone were reported. Participants who received oxycodone were reported.
Time Frame: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 36 | 37 | 35 | 37 | 36
ng*hr/mL/mg | 9.079 (2.7120) | 9.085 (2.3977) | 10.88 (2.9327) | 8.718 (2.4635) | 9.018 (2.6095)

49. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 3 - 7 days following last study drug administration. Symptoms of withdrawal following naloxone administration (naloxone challenge phase) were not collected as adverse events unless they met the criteria for an SAE. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Screening up to 28 days after last study drug administration (Day 29)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Naloxone: Naloxone HCl 0.2 mg intravenously followed by additional 0.6 mg naloxone HCl intravenously, each dose followed by an assessment for signs and symptoms of opioid withdrawal in naloxone challenge phase.
- Oxycodone HCl 40 mg: Single dose of oxycodone HCl 40 mg crushed tablet solution orally on either of 2 days in drug discrimination phase.
- Placebo Oxycodone HCl: Single dose of placebo matched to oxycodone HCl crushed tablet solution orally on either of 2 days in drug discrimination phase.
- Placebo: Single dose of matching placebo orally in either of the first to sixth intervention periods.
Arm/Group | Naloxone | Oxycodone HCl 40 mg | Placebo Oxycodone HCl | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 75 | 72 | 69 | 37 | 36 | 37 | 38 | 37 | 36
participants
  AEs | 5 | 70 | 14 | 12 | 29 | 37 | 27 | 34 | 36
  SAEs | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in Vital Sign Examinations
Description: Vital signs assessment included measurement of heart rate, systolic and diastolic blood pressures, respiratory rate and oral temperature. Criteria for clinically significant change in any vital sign examination was based on investigator's discretion.
Time Frame: Screening up to 7 days following last study drug administration (Day 8)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Naloxone | Oxycodone HCl 40 mg | Placebo Oxycodone HCl | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg
Number analyzed (Participants) | 75 | 72 | 69 | 37 | 36 | 37 | 38 | 37 | 36
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

51. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in End Tidal Carbon Dioxide (EtCO2)
Description: End-tidal carbon dioxide concentration in the expired air (EtCO2) was monitored using capnography in a sitting position. Criteria for clinically significant change in EtCO2 was based on investigator's discretion.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5 hours post-dose in drug discrimination phase; pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 14, 24, 36 hours post-dose in intervention period
Population: Safety analysis set included all participants who received at least 1 dose of study drug. This outcome measure was not planned to be analyzed in "Naloxone Challenge Phase", as pre-specified in protocol.
Measure: Number; unit: participants
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg | Oxycodone HCl 40 mg | Placebo Oxycodone HCl
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32 | 72 | 69
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

52. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in Oxygen Saturation of Hemoglobin (SpO2)
Description: Oxygen saturation of hemoglobin in blood (SpO2) was monitored using pulse oximetry continuously for 5 hours following dosing in the drug discrimination phase and continuously for 12 hours following dosing in the treatment phase, or longer at the discretion of the investigator. Individual measurements was collected in a sitting position. If SpO2 fall below 90 percent (%), the investigator might had administered oxygen via nasal cannula at a flow rate sufficient to maintain the SpO2 greater than or equal to 90%. Participants with fall in SpO2 below 90% were reported.
Time Frame: pre-dose up to 5 hours in drug discrimination phase; pre-dose up to 12 hours in intervention period
Population: as for outcome 51
Measure: Number; unit: participants
Arm/Group | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 mg- C | OXY 60 mg | Oxycodone HCl 40 mg | Placebo Oxycodone HCl
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32 | 72 | 69
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration (Day 29)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- ALO-02 60 Mg-C: Single dose of ALO-02 60 mg/7.2 mg crushed capsule (ALO-02 60 mg-C) solution orally in either of the first to sixth intervention periods.
Arm/Group | Naloxone | Oxycodone HCl 40 mg | Placebo | ALO-02 40 Mg-C | OXY 40 mg | ALO-02 60 Mg-I | ALO-02 60 Mg-C | OXY 60 mg | Placebo Oxycodone HCl
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/72 | 0/37 | 0/36 | 0/37 | 0/38 | 0/37 | 0/36 | 0/69
Other Adverse Events (participants affected / at risk) | 1/75 | 70/72 | 7/37 | 28/36 | 37/37 | 26/38 | 33/37 | 36/36 | 10/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxone (N=75) | Oxycodone HCl 40 mg (N=72) | Placebo (N=37) | ALO-02 40 Mg-C (N=36) | OXY 40 mg (N=37) | ALO-02 60 Mg-I (N=38) | ALO-02 60 Mg-C (N=37) | OXY 60 mg (N=36) | Placebo Oxycodone HCl (N=69)
Sinus arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxone (N=75) | Oxycodone HCl 40 mg (N=72) | Placebo (N=37) | ALO-02 40 Mg-C (N=36) | OXY 40 mg (N=37) | ALO-02 60 Mg-I (N=38) | ALO-02 60 Mg-C (N=37) | OXY 60 mg (N=36) | Placebo Oxycodone HCl (N=69)
Dry mouth (Gastrointestinal disorders) | 0 | 14 | 0 | 0 | 4 | 1 | 3 | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 13 | 3 | 4 | 6 | 5 | 6 | 7 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 2 | 2 | 1 | 4 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 2 | 5 | 4 | 4 | 4 | 3
Feeling hot (General disorders) | 0 | 11 | 1 | 2 | 5 | 1 | 7 | 2 | 1
Feeling of relaxation (General disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 10 | 0 | 6 | 8 | 7 | 7 | 10 | 2
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 4 | 7 | 5 | 4 | 0
Somnolence (Nervous system disorders) | 0 | 21 | 4 | 14 | 13 | 10 | 14 | 17 | 4
Euphoric mood (Psychiatric disorders) | 0 | 55 | 1 | 19 | 31 | 11 | 23 | 31 | 1
Hypervigilance (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 35 | 0 | 5 | 18 | 14 | 8 | 24 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 1 | 4 | 1 | 0 | 3 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.